CLINICAL TRIAL: NCT04400019
Title: Prevention of COVID19 Infection by the Administration of Hydroxychloroquine to Institutionalized Older People and Nursing Home Staff. Controlled Clinical Trial, Randomized Triple Blind by Clusters (PREVICHARM Study)
Brief Title: Prevention of COVID19 Infection in Nursing Homes by Chemoprophylaxis With Hydroxychloroquine (PREVICHARM)
Acronym: PREVICHARM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Collaborators: Instituto de Investigacion Biomedica de Malaga (Other); Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, JOSE MIGUEL MORALES ASENCIO, Professor of Research Methods and Evidence Based Health Care at University of Málaga (Spain), University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: COV20/00565
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Sars-CoV2; Coronavirus Infection; Prevention & Control; Nursing Home; Hydroxychloroquine
Keywords: clinical trial; Hydroxychloroquine; chemoprophylaxis; Sars-CoV2; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, triple-blind cluster study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The HCQ and the placebo will be manufactured by Laboratorios Rubio, blinded in similar containers for HCQ and placebo and will be stored in the pharmacy of the participating reference hospitals and will be distributed to the participating residences by the research technicians hired for the project.
  A record of doses delivered and monitoring of doses consumed will be carried out. The containers must be wrapped in a disposable protective cover, which can be removed before entering the residences, in order to minimize the accidental transmission of the virus through this route.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tracking control (No Intervention): According to the randomization process described, those nursing homes assigned to the control arm of the trial will receive the same treatment as those assigned to the intervention group, except for the medication, which will be a masked placebo.
  The study is triple blind, so neither the professionals who carry out the follow-up, nor the patients, nor the person in charge of analyzing the data, know to which group each nursing home belongs.
- Intervention (Experimental): The dose to be used as chemoprophylaxis will be 800mg of Hydroxychloroquine (HCQ) on the first day and 400mg during the subsequent four days. Participating subjects will be followed up at 6, 14 and 28 days.
  Interventions: Drug: Hydroxychloroquine Only Product in Oral Dose Form

INTERVENTIONS:
Drug: Hydroxychloroquine Only Product in Oral Dose Form — The dose to be used as chemoprophylaxis will be 800mg of HCQ on the first day and 400mg for the following four days.
  Arms: Intervention

SUMMARY:
Professionals and residents of nursing homes are one of the most vulnerable groups in this public health crisis of COVID-19, since they have the highest rate of positives for COVID-19, despite the restriction measures carried out, such as prohibition of family visits to these centers, the infection occurs by cross transmission with the care staff of the centers, or with other residents.

At the moment, there are no clinical trials to test the hypothesis that hydroxychloroquine is effective in coronavirus treatment. Although what has been observed is a better prognosis in infected patients, since this drug inhibits the replication of the virus and its expansion to other tissues.

This study is a clinical trial to test the effectiveness of hydroxychloroquine as a preventive drug for SARS-CoV-2 infection. This drug will be applied to 1050 people residing in nursing home care and 880 professionals who work in close contact with these people and who have not yet contracted the infection.

This project will be carried out in the territories of Madrid, Navarra, Aragon and Andalusia (Spain).

Hydroxychloroquine is a widely known drug that is used in two scenarios, against autoimmune diseases, such as lupus or rheumatoid arthritis, and as an antimalarial drug.

It is also intended to demonstrate that the presumed reduction in viral load that would be obtained with hydroxychloroquine prophylaxis, would have no effect in development of immunity against the virus. This fact can create a new paradigm for the de-escalation of the confinement to which the population has been subjected to stop the virus spread, allowing the development of general immunity in controlled populations until reaching total immunity.

In addition to testing the effect of this drug, a non-pharmacological intervention based on a safety record will be tested in the management of infection on nursing home, to assess its effectiveness in detecting risk areas or bad practices carried out in this vulnerable environment.

The study is led by researchers of the Institute of Biomedicine of Malaga (Spain), and has obtained a financing of 1,024,199 euros from Carlos III Health Institute (Spain).

The period of execution of the clinical trial is one year, and with this intervention, the intention is to reduce cross-infection in residents by a minimum threshold of 15%, as well as to decrease infection in the professionals.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness of hydroxychloroquine chemoprophylaxis in healthcare personnel and residents:

1. the incidence of secondary cases of SARS-CoV-2 infection in residents
2. the incidence of SARS-CoV-2 infection in the staff. To assess the effect of measures to promote infection control. Design: Controlled, randomized, triple-blind cluster multicentre trial. Subjects: Institutionalized older people and nursing homes staff in four Autonomous Communities.

Sample: 880 professionals, 1050 residents in 84 residences. They will be given 800mg of hydorxychloroquine the first day and 400mg in the subsequent four days. Nasopharyngeal exudate will be taken for baseline RT-PCR, and at six and 14 days after the adminsitration of hydroxychloroquine.

Mortality, compliance, safety, symptoms, and hospital admission will be evaluated secondarily.

The highest risk group for SARS-CoV-2 infection is that of people over 60 years of age, with cardiovascular disease, diabetes, COPD and immunosuppression, reaching up to 32% of those infected. But, in addition, the impact is especially insidious among institutionalized older people. The Spanish MInistry of Health has developed some regulations with measures to curb the impact in this context. WHO places institutionalized people as a very vulnerable group due to their permanent close contact with other people in the residence, the abundance of group activities, the presence of people with cognitive impairment and the need for help for their activities of daily living, which involves close physical contact with healthcare personnel. Even the interventions for preventing and controlling the infection could seriously affect the mental health and well-being of this vulnerable people, even if they do not contract the infection. In the province of Malaga (Spain), a checklist has been developed consisting of 13 items related to knowledge and compliance with the rules of prevention, self-protection, isolation and circuits, carried out by case management nurses. This instrument contains many of the WHO recommendations and may be an element that could make a difference in this context.

A significant proportion of those infected are known to have had close contact with probable or confirmed SARS-CoV-2 cases. In institutionalized people, the main source of contact (once family visits have been eliminated) is caused by cross-contamination with the care staff who provide direct care or other infected residents. In nursing homes, staff ratios are much more limited than in acute care hospitals (aggravated by the demand for professionals due to the epidemic). Furthermore, the possibility of isolation of infected patients is very limited: On average, residences only have 15% of their rooms prepared for isolation.

Among the various therapeutic strategies being tested, the use of hydroxychloroquine (HCQ) emerges as a viable option, albeit with limitations in the studies. This use has already been proposed for a long time due to its potential antiviral action, since it alkalinizes the cellular pH necessary for binding of the virus to the host cell and interferes with glycosylation of ECA2 receptors and blocks endosomatic transport of the virus. HCQ administered in a safe dose range is distributed throughout the body, including the lung parenchyma after oral administration, with few adverse effects. Compared to the antivirals under study for SARS-CoV-2 infection, it is much more feasible in real clinical practice conditions to access HCQ, a drug on which, in addition, there is enormous experience, its safety is well known, It is funded by the National Health System (NHS), it is cheap and accessible on the NHS. There are currently several clinical trials underway and a consensus has been developed that recommends their use in patients with SARS-CoV-2 pneumonia. Regarding the prophylactic use of HCQ, another trial in Spain has just started to use it in a "test and treat" strategy in patients among the general population, but it does not directly affect the institutionalized population. Our study aims to explore whether the administration of chemoprophylaxis in nursing homes is a protective strategy for both institutionalized people and the professionals themselves.

This is an controlled, randomized, triple-blind cluster study.The primary target population of the study consists of professionals who provide direct care in nursing homes (nursing assistants and nurses) and institutionalized older people.

The sampling frame will be integrated by the Communities of Andalusia, Madrid, Aragon and the Autonomous Community of Navarra. A conservative sample calculation has been designed, due to the current uncertainty regarding incidence. The incidence of Andalusia has been taken as the lower limit and the incidence provided in the study by Kimball et al. as an upper limit, and bearing in mind that many nursing homes are taking measures to isolate and relocate residents. To decrease the minimum infection rate in residents from 25% to 10% (delta = -0.15), with an alpha of 0.05, a power of 80%, assuming a minimum of 13 residents per cluster with a CCI of 0.1, with a replacement rate of losses of 25%, a total of 1050 residents would be necessary, with 7 clusters in each step, distributed in a total of 84 nursing homes. Regarding workers, taking the references from Andalusia and the study by McMichael et al. to decrease the minimum infection rate in professionals from 18% to 5% (delta = -0.13), with the same power parameters, assuming a minimum of 10 professionals per cluster with a CCI 0.1, and a replacement rate of 5% 880 professionals with the same number of clusters and nursing homes are required.

The PREVICHARM study was originally conceived at the end of March 2020 as a randomized clinical trial by stepped wedge clusters, since it was a methodological path that at that time allowed all participating subjects to receive the drug as chemoprophylaxis, in a staggered manner, without losing the comparison with a control group. After the evolution of the pandemic and the research around HCQ, the research team has considered the need to introduce some modifications in the design, to eliminate the staggering in the trial sequence, maintaining the design controlled and randomized by clusters, but, introducing an assignment of two parallel arms by triple blind to, on the one hand, have a totally blinded design that improves the robustness of the conclusions and, on the other, simplify the operationalization of the trial and thus further strengthen its feasibility. A criterion on the period of time necessary for inclusion has also been updated, reducing it to 8 days, in light of current knowledge on the predictive value of PCR in the course of infection in exposed patients.

The modifications do not affect the objectives, or hypotheses, or the outcomes, or the evaluation procedures thereof, or the follow-ups or the evaluation of the safety of the trial.

Variables: Sociodemographic, adjustment and control of confounders (Cluster, follow-up time, hours worked by each professional during the study, gradient of application of non-pharmacological measures); Primary endpoints: Number of secondary cases of SARS-CoV2 infection among residents, and SARS-CoV-2 infection in caregivers who provide direct care; Secondary endpoints: mortality, compliance with treatment, symptoms of SARS-CoV-2 infection, hospital admission of personnel and adverse events.

All the nursing homes in the province will be invited to participate and after randomization, the phased inclusion of residences will begin, requesting the consent of professionals to be included and proceeding to collect basal exudate and study variables. In the randomized nursing homes in each step as an intervention, the HCQ regimen will be provided and the nasopharyngeal exudate follow-up will be performed for RT-PCR at 6 and 14 days. In those in the control group step, an exudate will be collected on the same days than intervention group. Once enrolled, subjects will receive a double naso-oro-pharyngeal swab and will be provided blinded medication (HCQ or placebo, as appropriate) for the entire chemoprophylaxis cycle. Subsequently, smears will be taken again at 6 and 14 days. The sample collection procedure will be standardized through the protocol developed by the Ministry of Health and technicians will be trained in advance in its performance.

The technicians will go to each residence according to a cadence pre-established by the research team.

Adverse events will be monitored at each weekly visit using a standardized procedure (gastrointestinal disorders, appetite disturbances, hypoglycemia, weight loss, decreased visual acuity, photophobia, impaired visual accommodation with symptoms of blurred vision, deafness, tinnitus, and vertigo, muscle weakness, symptoms of liver and kidney disorders, neurological disorders). Serious and non-serious adverse events will be distinguished and will be notified by means of a standard procedure to the Research Ethics Committee, and to the Spanish Agency for Medicines and Health Products. An insurance policy has been contracted for risk coverage.

The study will comply with all the precepts of the Declaration of Helsinki and its subsequent revisions, as well as the Standards of Good Practice. Participants will be informed of the characteristics and purpose of the study and will be asked for informed consent in accordance with the regulations in force in Spain using the form and the corresponding information sheet. The study has been approved by the Malaga Provincial Research Ethics Committee and the Spanish Agency for Medicines and Health Products, as well as the participating institutions.

All the trial monitoring process and pharmacovigilance will be carried out by the Clinical Trial Units of the Spanish Clinical Research Network of the participating Centers.

Exploratory data analysis, bivariate analysis (chi square, Student t, ANOVA or their non-parametric equivalents in case of non-normality) will be performed and the main hypothesis will be tested using generalized linear binomial and Poisson models, also taking the cluster, as random effects factor, and time as a fixed factor. Intrasubject analyzes will be carried out using mixed generalized linear models. All the analyses will be performed by intention to treat, using multiple imputation models.

The total estimated duration is a maximum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized people in nurswing homes since the beginning of the COVID19 epidemic who do not have the infection present at the time of entering into the study.
* Healthcare professionals who provide direct care (nursing assistants and registered nurses) to institutionalized older people in nursing homes with confirmed cases of COVID19 during the past 8 days.
* Subjects that give their consent to participate in the study or that it be obtained from their representative / legal guardian.

Exclusion Criteria:

* Staff members who do not provide direct care to residents.
* Residents with active SARS-CoV-2 infection present, or with symptoms compatible with COVID19 confirmed by PCR test.
* Staff members with present or past SARS-CoV-2 infection, or with PCR-confirmed symptoms consistent with COVID19.
* History of QT interval prolongation or arrhythmias of any etiology.
* Presence of retinopathy of any etiology, changes in acuity or visual field.
* Severe hearing loss (requires the use of hearing aids).
* Structural heart disease.
* History of non-structural heart failure, ischemic heart disease, SCASEST, or SCACEST
* Chronic liver disease.
* Alcoholism.
* Epilepsy.
* For the participating professionals, pregnancy or suspected pregnancy (if they are planning pregnancy, or in fertilizer treatment, they must abandon the study).
* Subjects with known HDQ hypersensitivity.
* Subjects diagnosed with G6PDH deficiency.
* Taking other medicines that prolong QT: domperidone, ondansetron, cilostazol, antiarrhythmics (procainamide, amiodarone, flecainide, sotalol), macrolides (azithromycin, clarithromycin, erythromycin), quinolones (ciprofloxacin,), moxofloxacin,) neuroleptics (haloperidol, chlorpromazine, pimozide), antidepressants (citalopram, escitalopram), sulpiride, anticholinesterase drugs (donepezil)
* Denial to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1930 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of secondary cases of SARS-CoV2 infection among residents at six days | This outcome will be evaluated at six days from the administration of chemoprophylaxis with hydroxychloroquine
  Discrete quantitative variable. Residents with active viral load (diagnosed by polymerase chain reaction test) will be considered infected.
Number of secondary cases of SARS-CoV2 infection among residents at 14 days | This outcome will be evaluated at 14 days from the administration of chemoprophylaxis with hydroxychloroquine
  Discrete quantitative variable. Residents with active viral load (diagnosed by polymerase chain reaction test) will be considered infected.
Number of secondary cases of SARS-CoV2 infection among residents at 28 days | This outcome will be evaluated at 28 days from the administration of chemoprophylaxis with hydroxychloroquine
  Discrete quantitative variable. Residents with active viral load (diagnosed by polymerase chain reaction test) will be considered infected.
SARS-CoV-2 infection in nursing home staff who provide direct care at six days | This outcome will be evaluated at six days from the administration of chemoprophylaxis with hydroxychloroquine
  Dichotomous categorical variable
SARS-CoV-2 infection in nursing home staff who provide direct care at 14 days | This outcome will be evaluated at 14 days from the administration of chemoprophylaxis with hydroxychloroquine
  Dichotomous categorical variable
SARS-CoV-2 infection in nursing home staff who provide direct care at 28 days | This outcome will be evaluated at 28 days from the administration of chemoprophylaxis with hydroxychloroquine
  Dichotomous categorical variable

SECONDARY OUTCOMES:
Mortality | This outcome will be evaluated at 28 days from the administration of chemoprophylaxis with hydroxychloroquine
  Dichotomous qualitative variable (1: Death 0: Survival)
Compliance with treatment | It will be evaluated during the five days that the chemoprophylaxis with hydorxychloroquine is administered
  Continous variable. It will be evaluated with the AIDS Clinical Trials Group method: investigation of medications not taken in a period of 4 days prior to the interview)% adherence = (total prescribed galenic units for that period-total units not taken) / total prescribed galenic units for that period
Symptoms of SARS-CoV-2 infection at six days | This outcome will be evaluated at 6 days from the administration of chemoprophylaxis with hydroxychloroquine
  Dichotomous categorical variable. The participant presents symptoms compatible with SARS-CoV-2 infection. High temperature, cephalea, dyspnea,diarrhea, vomiting, arthro-myalgia, pharynx pain, abdominal pain, anosmia, cough.
Symptoms of SARS-CoV-2 infection at 14 days | This outcome will be evaluated at 14 days from the administration of chemoprophylaxis with hydroxychloroquine
  Dichotomous categorical variable. The participant presents symptoms compatible with SARS-CoV-2 infection. High temperature, cephalea, dyspnea,diarrhea, vomiting, arthro-myalgia, pharynx pain, abdominal pain, anosmia, cough.
Symptoms of SARS-CoV-2 infection at 28 days | This outcome will be evaluated at 28 days from the administration of chemoprophylaxis with hydroxychloroquine
  Dichotomous categorical variable. The participant presents symptoms compatible with SARS-CoV-2 infection. High temperature, cephalea, dyspnea,diarrhea, vomiting, arthro-myalgia, pharynx pain, abdominal pain, anosmia, cough.
Hospitalization | This outcome will be evaluated at 28 days from the administration of chemoprophylaxis with hydroxychloroquine
  Dichotomous categorical variable. Participant requires hospital admission attributable to SARS-CoV-2 infection
Adverse events at six days | This outcome will be evaluated at six days from the administration of chemoprophylaxis with hydroxychloroquine
  Polycotomic categorical variable. Collected by clinical interview and also monitored simultaneously by external trial monitors
Adverse events at 14 days | This outcome will be evaluated at 14 days from the administration of chemoprophylaxis with hydroxychloroquine
  Polycotomic categorical variable. Collected by clinical interview and also monitored simultaneously by external trial monitors
Adverse events at 28 days | This outcome will be evaluated at 28 days from the administration of chemoprophylaxis with hydroxychloroquine
  Polycotomic categorical variable. Collected by clinical interview and also monitored simultaneously by external trial monitors

CONTACTS AND LOCATIONS:
Overall Officials: José M Morales-Asencio, PhD, Principal Investigator — University of Malaga; Malaga, Spain.; Ricardo Gómez-Huelgas, PhD, Principal Investigator — Hospital Regional de Malaga; Juan C Morilla-Herrera, PhD, Principal Investigator — Distrito de Atención Primaria Málaga-Valle del Guadalhorce

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganyani T, Kremer C, Chen D, Torneri A, Faes C, Wallinga J, Hens N. Estimating the generation interval for coronavirus disease (COVID-19) based on symptom onset data, March 2020. Euro Surveill. 2020 Apr;25(17):2000257. doi: 10.2807/1560-7917.ES.2020.25.17.2000257. PMID 32372755
- [Background] Pan Y, Zhang D, Yang P, Poon LLM, Wang Q. Viral load of SARS-CoV-2 in clinical samples. Lancet Infect Dis. 2020 Apr;20(4):411-412. doi: 10.1016/S1473-3099(20)30113-4. Epub 2020 Feb 24. No abstract available. PMID 32105638
- [Background] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Background] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Yan Y, Zou Z, Sun Y, Li X, Xu KF, Wei Y, Jin N, Jiang C. Anti-malaria drug chloroquine is highly effective in treating avian influenza A H5N1 virus infection in an animal model. Cell Res. 2013 Feb;23(2):300-2. doi: 10.1038/cr.2012.165. Epub 2012 Dec 4. No abstract available. PMID 23208422
- [Background] Savarino A, Di Trani L, Donatelli I, Cauda R, Cassone A. New insights into the antiviral effects of chloroquine. Lancet Infect Dis. 2006 Feb;6(2):67-9. doi: 10.1016/S1473-3099(06)70361-9. No abstract available. PMID 16439323
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Shipman WD, Vernice NA, Demetres M, Jorizzo JL. An update on the use of hydroxychloroquine in cutaneous lupus erythematosus: A systematic review. J Am Acad Dermatol. 2020 Mar;82(3):709-722. doi: 10.1016/j.jaad.2019.07.027. Epub 2019 Jul 13. PMID 31306730
- [Background] multicenter collaboration group of Department of Science and Technology of Guangdong Province and Health Commission of Guangdong Province for chloroquine in the treatment of novel coronavirus pneumonia. [Expert consensus on chloroquine phosphate for the treatment of novel coronavirus pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):185-188. doi: 10.3760/cma.j.issn.1001-0939.2020.03.009. Chinese. PMID 32164085
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Background] McMichael TM, Currie DW, Clark S, Pogosjans S, Kay M, Schwartz NG, Lewis J, Baer A, Kawakami V, Lukoff MD, Ferro J, Brostrom-Smith C, Rea TD, Sayre MR, Riedo FX, Russell D, Hiatt B, Montgomery P, Rao AK, Chow EJ, Tobolowsky F, Hughes MJ, Bardossy AC, Oakley LP, Jacobs JR, Stone ND, Reddy SC, Jernigan JA, Honein MA, Clark TA, Duchin JS; Public Health-Seattle and King County, EvergreenHealth, and CDC COVID-19 Investigation Team. Epidemiology of Covid-19 in a Long-Term Care Facility in King County, Washington. N Engl J Med. 2020 May 21;382(21):2005-2011. doi: 10.1056/NEJMoa2005412. Epub 2020 Mar 27. PMID 32220208
- [Background] Kimball A, Hatfield KM, Arons M, James A, Taylor J, Spicer K, Bardossy AC, Oakley LP, Tanwar S, Chisty Z, Bell JM, Methner M, Harney J, Jacobs JR, Carlson CM, McLaughlin HP, Stone N, Clark S, Brostrom-Smith C, Page LC, Kay M, Lewis J, Russell D, Hiatt B, Gant J, Duchin JS, Clark TA, Honein MA, Reddy SC, Jernigan JA; Public Health - Seattle & King County; CDC COVID-19 Investigation Team. Asymptomatic and Presymptomatic SARS-CoV-2 Infections in Residents of a Long-Term Care Skilled Nursing Facility - King County, Washington, March 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 3;69(13):377-381. doi: 10.15585/mmwr.mm6913e1. PMID 32240128
- [Background] Quagliarello V, Ginter S, Han L, Van Ness P, Allore H, Tinetti M. Modifiable risk factors for nursing home-acquired pneumonia. Clin Infect Dis. 2005 Jan 1;40(1):1-6. doi: 10.1086/426023. Epub 2004 Dec 1. PMID 15614684
- [Background] Chesney MA, Ickovics JR, Chambers DB, Gifford AL, Neidig J, Zwickl B, Wu AW. Self-reported adherence to antiretroviral medications among participants in HIV clinical trials: the AACTG adherence instruments. Patient Care Committee & Adherence Working Group of the Outcomes Committee of the Adult AIDS Clinical Trials Group (AACTG). AIDS Care. 2000 Jun;12(3):255-66. doi: 10.1080/09540120050042891. PMID 10928201
- [Background] Pagarolas AA, Sune TP. [Microbiological diagnosis of viral respiratory infections in the adult patient]. Enferm Infecc Microbiol Clin. 2014 Feb;32 Suppl 1:51-6. doi: 10.1016/S0213-005X(14)70150-8. Spanish. PMID 24630584
- [Background] Kalil AC. Treating COVID-19-Off-Label Drug Use, Compassionate Use, and Randomized Clinical Trials During Pandemics. JAMA. 2020 May 19;323(19):1897-1898. doi: 10.1001/jama.2020.4742. No abstract available. PMID 32208486
- See also: Sociedad Española de Geriatría y Gerontología. Colaboración servicios de geriatría hospitalarios - hospitales de media estancia - residencias de mayores y centros sociosanitarios. 2020 — https://www.segg.es/media/descargas/pautas-SEGG-covid-19.pdf
- See also: Mitja O. Antiviral Treatment of COVID-19 Confirmed Cases and Ring Chloroquine Chemoprevention in Close Contacts: a Cluster Randomized Clinical Trial. 2020 [cited 2020 Mar 22]. (Clinical Trials.gov). Report No.: NCT04304053. — https://www.clinicaltrialsregister.eu/ctr-search/trial/2020-000890-25/FR